CLINICAL TRIAL: NCT00147771
Title: Evaluation of the Efficacy and Safety of the Imiquimod 5% Topical Cream in Plaque Morphea: A Prospective, Multiple Baseline, Open Label Pilot Study
Brief Title: Imiquimod in Children With Plaque Morphea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elena Pope, Head, Section of Dermatology, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000007595
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Scleroderma, Localized
Keywords: localized scleroderma; morphea; imiquimod; pediatrics
MeSH Terms: conditions — Scleroderma, Localized | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Imiquimod 5% cream — Treatment will last for 36 weeks. Patients will be instructed to apply Imiquimod three times per week for 4 weeks. If no local side effects are noted at the 4 week- follow-up visit, the frequency of the application will be increased to 5 weekly applications.

SUMMARY:
Morphea is very hard to treat. In a small number of adult patients, Imiquimod has proven to be beneficial in decreasing the thickness of the morphea plaques , while improving their appearance. There are no studies to date proving its safety and efficacy in children with this disease. We propose to conduct a pilot study to assess to potential efficacy and relative safety of Imiquimod in children with plaque morphea.

DETAILED DESCRIPTION:
Design: Prospective, open label, pilot study

Settings: The Hospital for Sick Children, Specialized Morphea Clinic

Study population:

* Children 6-18 years of age
* Plaque morphea measuring less than 10 cm2 in diameter ( for children with multiple lesions, only one will be treated)

Intervention: Topical imiquimod applied 3-5 times a week for 6 months

Outcome measures: Decrease in the thickness of the skin by clinical scores and ultrasonography

Duration of the study: 12 months ( 2 baseline visits, 1 intervention visit, 5 follow-up visits)

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis 6 to 18 years of age
* Morphea plaques
* Female subjects of childbearing potential must have a negative urine pregnancy test
* Signed consent/assent form

Exclusion criteria:

* Children who received topical corticosteroids, tacrolimus, vitamin D derivatives (calcipotriol, calcipotriol-betamethasone dipropionate) to the affected area in the previous four weeks
* Children who were previously treated with Imiquimod on the affected areas
* Children with no demonstrable ultrasonographic changes at the baseline evaluation
* Children with evidence of skin breakdown on the proposed area to be treated at the time of enrollment due to potential increased absorption of the medication through impaired skin barrier
* Female subjects of childbearing potential who do not agree to practice effective birth control methods for the duration of the study
* Children who are/were (in the past 6 months) treated with systemic medications such as methotrexate and/or systemic corticosteroids
* Co-morbidities: systemic sclerosis, juvenile rheumatoid arthritis, other systemic diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Percent improvement in the thickness of the skin | 4 weeks, 12 weeks, 24 weeks, 36 weeks, and 48 weeks

SECONDARY OUTCOMES:
Frequency of side-effects | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada